CLINICAL TRIAL: NCT00078143
Title: Motivational Enhancement Therapy (MET) to Improve Treatment Utilization in Pregnant Substance Users
Brief Title: Motivational Enhancement Therapy to Improve Treatment Utilization in Pregnant Substance Users - 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Responsible Party: Theresa Winhusen, Ph.D., University of Cincinnati
Organization: National Institute on Drug Abuse (NIDA) (NIH)
Purpose: Treatment
Other Study IDs: NIDA-CTN-0013-1
Record Dates: First submitted 2004-02-19; First posted 2004-02-23 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2016-10

CONDITIONS: Substance-Related Disorders
Keywords: behavioral intervention
MeSH Terms: conditions — Substance-Related Disorders | interventions — Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Behavior Therapy

SUMMARY:
The purpose of this study is to compare Motivational Enhancement Therapy (MET) with standard drug abuse treatment among pregnant women.

ELIGIBILITY:
Inclusion Criteria:

* Pregnancy <30 weeks
* Have not attended drug treatment in past 28 days
* Not needing residential treatment (except detox)
* Not at risk for suicide/homicide
* Have no pending legal charges (except drug treatment)

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2003-10; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Treatment Utilization
Substance Abuse

CONTACTS AND LOCATIONS:
Overall Officials: Theresa Winhusen, Ph.D., Principal Investigator — University of Cincinnati
Locations (6):
- United States (6):
  - Midtown Community Mental Health Center, Indianapolis, Indiana
  - Jefferson Alcohol & Drug Abuse Center, Louisville, Kentucky
  - Eleonore Hutzel Recovery Center, Detroit, Michigan
  - Milagro Clinic, Albuquerque, New Mexico
  - Milagro, Albuquerque, New Mexico
  - Coastal Horizons Center, Inc., Wilmington, North Carolina

REFERENCES:
- [Derived] Osterman R, Lewis D, Winhusen T. Efficacy of motivational enhancement therapy to decrease alcohol and illicit-drug use in pregnant substance users reporting baseline alcohol use. J Subst Abuse Treat. 2017 Jun;77:150-155. doi: 10.1016/j.jsat.2017.02.003. Epub 2017 Feb 21. PMID 28254158
- [Derived] Winhusen T, Lewis D. Cigarette smoking in pregnant substance users: Association with substance use and desire to quit. J Addict Dis. 2017 Jan-Mar;36(1):88-91. doi: 10.1080/10550887.2016.1254992. Epub 2016 Nov 1. PMID 27802114